CLINICAL TRIAL: NCT02286999
Title: A Parallel-group, Randomized, Placebo-controlled Ascending Dose Phase I Study Protocol for Dietary Supplementation With Bifidobacterium Longum Subsp. Infantis (B. Infantis) in Healthy Breastfed Infants
Brief Title: Probiotic Supplementation in Breastfed Newborn Infants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study did not open for enrollment.
Sponsor: Emanual Maverakis, MD (Other)
Responsible Party: Sponsor-Investigator, Emanual Maverakis, MD, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 651698
Record Dates: First submitted 2014-10-23; First posted 2014-11-10 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Atopic Dermatitis; Food Allergies
MeSH Terms: conditions — Dermatitis, Atopic; Food Hypersensitivity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- B.infantis (Experimental): Infants in the experimental arm will have two doses of the probiotic Bifidobacterium longum subsp. infantis (B. infantis) on Day 7 and Day 14 of life.
  Interventions: Drug: B. infantis
- Placebo (Placebo Comparator): Infants in the experimental arm will have two doses of placebo (powdered maltodextrin) on Day 7 and Day 14 of life.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: B. infantis — Infants in the intervention group will receive two doses of B. infantis on Day 7 and Day 14 of life, while infants in the placebo group will be dosed with placebo on Day 7 and Day 14
  Other Names: Probiotic
  Arms: B.infantis
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the dose of a probiotic supplement (Bifidobacterium longum subsp. infantis) required to achieve predominant gut colonization in healthy newborn, breastfed infants. The study will also examine whether supplementation with this probiotic can reduce the chance of developing eczema and food allergies in enrolled infants.

DETAILED DESCRIPTION:
The proposed phase I clinical trial is a parallel-group, placebo-controlled, randomized, double-blind ascending dose study of dietary supplementation with Bifidobacterium longum subsp. infantis (B. infantis) in healthy breastfed infants to evaluate its safety as well as determine the pharmacologically effective dose (ED) of B. infantis producing at least 50% gut colonization at six weeks of age. Infants will be enrolled sequentially in groups of five (three randomized to receive B. infantis and two to receive placebo). For each group, infants will be dosed with B. infantis or placebo on day 7 and day 14 of life. A calculated Maximally Recommended Starting Dose (MRSD) will be used to initiate the dose escalation and is defined below. Every two weeks, an additional group of five infants (randomized 3:2 to B. infantis and placebo) will be enrolled to receive progressively higher doses of B. infantis. Calculation of the appropriate dose escalation will be performed using a modified Fibonacci series as described below in an effort to identify the ED of B. infantis.

After the ED of B. infantis has been identified (defined as the dose capable of producing 50% gut colonization by six weeks of age) two additional sequential dose escalations will be performed. The purpose of the final two dose escalations is to determine if successively higher doses of B. infantis result in increased gut colonization or barrier protection; or, alternatively, if a Maximum Effective Dose (MaxED) for B. infantis exists above which there is no further increase in gut colonization or barrier protection. Following the final dose escalation, Hanley's Rule of Three will be applied in order to determine if lower-frequency adverse events are caused by B. infantis. Hanley's Rule of Three states that in order to identify any adverse events occurring at a frequency of 1:10 or greater with a 95% confidence interval, at least 30 subjects must be enrolled.

Study visits will be scheduled for weeks 1, 2, 6, 24, 36, 52 and 78. Parents will complete surveys at each study visit to monitor the infants for potential adverse events associated with probiotic administration including feeding intolerance, fevers, or bowel irregularities including constipation and diarrhea.

Stool samples will be collected twice weekly for the first six weeks of life then once weekly at weeks 24, 36, 52 and 78. Stool samples will be analyzed to determine the relative abundance of B. infantis over time, and the overall diversity of the gut microbiota with and without B. infantis supplementation. Stool will also be analyzed for milk oligosaccharides to verify consumption of breast milk and to correlate proportion of human milk oligosaccharides and free sugar monomers seen in the infant stool at various levels of B. infantis colonization.

At each study visit, infants will receive a full skin examination to evaluate for signs of atopic dermatitis (AD). The Infant Dermatitis Quality of Life Index (IDQOLI) will be administered to parents at each study visit to screen for possible signs of AD such as infant irritability, skin rashes and hypersensitivity. If AD is present, the Scoring Atopic Dermatitis (SCORAD) grading system will be used to assess severity. Urine samples will be collected at each study visit to measure levels of fatty acid binding proteins (FABPs) and glutathione-S-transferase (alpha-GST), which are non-invasive markers of gastrointestinal permeability that may indicate the presence of food allergies. Blood will be collected via finger or heel stick at weeks 6 and 52 for immune phenotyping (including measuring inflammatory cytokines and food-specific IgEs). In addition, levels of serum fatty acid binding proteins (FABPs) and glutathione-S-transferase (alpha-GST) will be measured as markers of gastrointestinal permeability and potential food allergy. Parents will also complete surveys at each study visit to monitor the infants for potential adverse events associated with probiotic administration including feeding intolerance, fevers, or bowel irregularities including constipation and diarrhea.

Entry into the study requires the intent to breastfeed exclusively for a minimum of six months. If mothers decide to discontinue breastfeeding during the study, the investigators will note that in the infant's chart and obtain an additional series of weekly stool samples for six weeks after discontinuation of breastfeeding. The purpose of this additional stool sample collection is to determine if discontinuation of breastfeeding has an impact on the level of existing B. infantis colonization in the infant gut.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn infants between 1 and 7 days old with intent to be exclusively breastfed for a minimum of six (6) months

Exclusion Criteria:

* Infants given dietary supplementation, including other probiotics.
* Infants born prior to 34 weeks gestation.
* Infants below 10th percentile for body weight.
* Postnatal use of antibiotics (oral, intramuscular or intravenous) by either the mother or the infant. Of note, prenatal maternal Group B streptococcus prophylaxis is not a criterion for study exclusion.
* Family history of immunodeficiency syndrome(s).
* Infants with signs of a clinically apparent underlying immunodeficiency.
* Intent to use non-breast milk infant formula for feeding during the first six months.
* History of GI tract abnormality or infection.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Pharmacologically effective dose (ED) of B. infantis | Two years
  The primary endpoint of the study is identification of a pharmacologically effective dose of B. infantis required to produce predominant (>50%) gut colonization at six weeks of age
Safety of Probiotic Supplementation, as assessed by frequency of adverse events | 2 years
  An additional primary endpoint is to determine the safety of B. infantis supplementation in immunocompetent, full-term infants. Any adverse events including fever 102°F or higher, abdominal pain or colic, blood or pus in the stool, diarrhea or vomiting will be documented and dosing adjusted accordingly

SECONDARY OUTCOMES:
Milk Oligosaccharide Consumption | 2 years
  All stool samples will also be analyzed for the presence of oligosaccharides unique to breast milk and for the presence of free saccharide monomers, which are products of their incomplete digestion. B. infantis abundance will be correlated to these values.
Stool Microbiota Composition | 2 years
  In addition to determining the percent composition of B. infantis in infant stool samples, numerous other measures such as microbiota diversity and rate of B. infantis decline following cessation of breast feeding will also be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Emanual Maverakis, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Awasthi S, Wilken R, Patel F, German JB, Mills DA, Lebrilla CB, Kim K, Freeman SL, Smilowitz JT, Armstrong AW, Maverakis E. Dietary supplementation with Bifidobacterium longum subsp. infantis (B. infantis) in healthy breastfed infants: study protocol for a randomised controlled trial. Trials. 2016 Jul 22;17(1):340. doi: 10.1186/s13063-016-1467-1. PMID 27449926